CLINICAL TRIAL: NCT04749745
Title: Effects of Single-dose L-theanine on Motor Cortex Excitability in Healthy Subjects: A Double-blinded, Randomized Order, Cross-over Paired-Pulse Transcranial Magnetic Stimulation Study
Brief Title: Effects of L-theanine on Motor Cortex Excitability in Healthy Subjects: A Paired-Pulse TMS Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 202006-003
Record Dates: First submitted 2021-01-27; First posted 2021-02-11 (Actual); Results first posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-08

CONDITIONS: Cortical Excitability; Psychiatric Disorder
Keywords: L-theanine; Cortical Excitability; NMDA; GABA; Paired-Pulse TMS
MeSH Terms: conditions — Mental Disorders | interventions — theanine

STUDY DESIGN:
Intervention Model Description: This is a pilot study, investigating the effects of single dose L-theanine in Healthy subjects, to further assess the validity and feasibility to study this compound in patient population.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-Theanine (Active Comparator): Subject will receive 400mg single dose of L-theanine, by oral ingestion with water. The capsules are prepared and dispensed by hospital pharmacy, with the investigator and participant both blinded.
  Interventions: Drug: L-theanine; Drug: Placebo
- Placebo (Placebo Comparator): Subject will receive 400mg single dose of matching Placebo, by oral ingestion with water. The capsules are prepared and dispensed by hospital pharmacy, with the investigator and participant both blinded.
  Interventions: Drug: L-theanine; Drug: Placebo

INTERVENTIONS:
Drug: L-theanine — The subject will receive paired-pulse TMS (ppTMS) procedure before and 30min after taking the drug orally, to assess motor cortex excitability, measured by surface electromyogram (EMG). The ppTMS procedure is administered by a TMS stimulator controlled a program software named Signal. The coil of the stimulator is placed above the scalp where the stimulation would activate the left primary motor cortex region that controls the right thumb. When a pulse stimulation is delivered by the coil, the EMG over a thumb muscle (abductor pollicis brevis) will record a motor-evoked potential on the tracing. Cross-over with placebo in two separate sessions at least 72 hours apart.
Drug: Placebo — The subject will receive paired-pulse TMS (ppTMS) procedure before and 30min after taking the drug orally, to assess motor cortex excitability, measured by surface electromyogram (EMG). The ppTMS procedure is administered by a TMS stimulator controlled a program software named Signal. The coil of the stimulator is placed above the scalp where the stimulation would activate the left primary motor cortex region that controls the right thumb. When a pulse stimulation is delivered by the coil, the EMG over a thumb muscle (abductor pollicis brevis) will record a motor-evoked potential on the tracing. Cross-over with L-theanine in two separate sessions at least 72 hours apart.

SUMMARY:
Major depressive disorder (MDD) is a serious mental illness and the leading cause of disability worldwide. New pharmacotherapeutic agents with complementary neurobiological mechanism and better side effect profile are of great needs. In addition to the monoamine system, the glutamatergic system plays a crucial role in MDD.

L-theanine (N5-ethyl-L-glutamine) is the primary psychoactive component uniquely in green tea. Preclinical studies have demonstrated anti-depressant effect of L-theanine in rodents and provided evidences for its pharmacological properties of N-methyl-D-aspartate (NMDA) and gamma-aminobutyric acid (GABA) agonism. Yet these effects have not been proven in humans. Only one open-label clinical trial has studied and supported antidepressant effects of L-theanine in MDD patients. We propose using pair-pulse transcranial magnetic stimulation (ppTMS) to probe how L-theanine may manipulate the glutamatergic and GABA systems in the frontal region by changing cortical excitability first in healthy subjects. We plan to investigate the neurobiological effects of L-theanine in healthy subjects first.

Granted that the first phase pilot trial provides neurophysiological evidence of L-theanine on motor cortex excitability in human subjects, next phases of studies on L-theanine in MDD patients cortical excitability could be justified.

DETAILED DESCRIPTION:
Background and Significance:

Major depressive disorder (MDD) is a serious mental illness and the leading cause of disability worldwide. Although many antidepressants acting on synaptic monoamine levels have been used as the first-line drug treatment for MDD, around one third of MDD are pharmacologically resistant. Side effects of these medications impose additional hardship on adherence and further affect treatment outcome. New pharmacotherapeutic agents with complementary neurobiological mechanism and better side effect profile are of great needs. In addition to the monoamine system, the glutamatergic system plays a crucial role in MDD.

L-theanine (N5-ethyl-L-glutamine) is the primary psychoactive component uniquely in green tea. Epidemiological studies support that green tea consumption is an independent factor associated with lower prevalence of depression. Preclinical studies have demonstrated anti- depressant effect of L-theanine in rodents and provided evidences for its pharmacological properties of N-methyl-D-aspartate (NMDA) and gamma-aminobutyric acid (GABA) agonism. Yet these effects have not been proven in humans. Only one open-label clinical trial has studied and supported antidepressant effects of L-theanine in MDD patients. We propose using pair-pulse transcranial magnetic stimulation (ppTMS) to probe how L-theanine may manipulate the glutamatergic and GABA systems in the frontal region by changing cortical excitability first in healthy subjects. ppTMS is a well-established technique to investigate frontal motor cortical excitability mediated by the inter-neuron NMDA and GABA receptors. Specific changes of ppTMS measures, including impaired short-term and long-term intracortical inhibition (SICI, mediated by GABA-A receptor; LICI, mediated by GABA-B receptor) and intracortical facilitation (ICF, mediated by NMDA receptor), have been demonstrated in MDD. Using this technique, we plan to investigate the neurobiological effects of L-theanine in healthy subjects first.

Granted that the first phase pilot trial provides neurophysiological evidence of L-theanine on motor cortex excitability in human subjects, next phases of studies on L-theanine in MDD patients cortical excitability could be justified. This will lay foundation for further exploration of L-theanine's potential as an augmenting agent for MDD in a placebo- controlled design.

Aims and Hypothesis:

Given the potential NMDA and GABA agonistic effects of L-theanine, we hypothesize that it increases intracortical inhibition and facilitation through enhancement of NMDA- and GABA-receptor mediated neurotransmission, in healthy subjects (N=10 to complete study).

Study Procedures:

Double-blinded, Randomized-order, Cross-over placebo-controlled to evaluate acute effect of single-dose L-theanine on motor cortex excitability by ppTMS in 10 healthy subjects.

Dose of L-theanine or placebo is 400mg. At baseline, subjects will be randomized to L- theanine or placebo group, then receive ppTMS protocol before drug administration. The ppTMS protocol is repeated after 30min of administration. Then subjects will return to clinic after 1 week free of any medications and repeat the above protocol with the second drug condition. Visual analog scale will be used to evaluate psychosomatic symptoms and wellbeing of the subjects pre- and post-each drug administration.

Data Analytic Plan:

Wilcoxon test will be used to compare the baseline-to-post-drug means of SICI, LICI and ICF measures. Prespecified covariates include age, sex, handedness, level of fatigue will be analyzed in linear regression model. The time-condition relationship with continuous dependent variables of ICI and ICF values will be evaluated by Mixed Effect Model. Two- sided P value < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, aged between 18 and 65 years old;
2. Able to read/speak English and give informed consent
3. No current or history of Axis I psychiatric disorders by DSM-5.
4. Free of psychotropic medication use

Exclusion Criteria:

1. History of significant acute or chronic neurological or medical disorder or condition that increases risk for seizure with TMS;
2. History of alcohol use disorder, nicotine dependence, adjustment disorder;
3. History of allergic reactions to L-theanine or green tea;
4. Pregnancy;
5. Unable/unwilling to abstain from nutraceutical supplements and psychotropic agents during participation in the study
6. Unable/ unwillingness to refrain from recreational substance use (e.g. alcohol or marijuana) during participation in the study;
7. Meet criteria for exclusion from TMS or MRI procedures, including intracranial metal implants or nonremovable ferromagnetic items in the head/neck.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Carpenter, MD, Principal Investigator — Brown University-Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
To protect subject confidential information.

REFERENCES:
- [Background] Vuong QV, Bowyer MC, Roach PD. L-Theanine: properties, synthesis and isolation from tea. J Sci Food Agric. 2011 Aug 30;91(11):1931-9. doi: 10.1002/jsfa.4373. Epub 2011 Mar 29. PMID 21735448
- [Background] Kim J, Kim J. Green Tea, Coffee, and Caffeine Consumption Are Inversely Associated with Self-Report Lifetime Depression in the Korean Population. Nutrients. 2018 Sep 1;10(9):1201. doi: 10.3390/nu10091201. PMID 30200434
- [Background] Hintikka J, Tolmunen T, Honkalampi K, Haatainen K, Koivumaa-Honkanen H, Tanskanen A, Viinamaki H. Daily tea drinking is associated with a low level of depressive symptoms in the Finnish general population. Eur J Epidemiol. 2005;20(4):359-63. doi: 10.1007/s10654-005-0148-2. PMID 15971509
- [Background] Hozawa A, Kuriyama S, Nakaya N, Ohmori-Matsuda K, Kakizaki M, Sone T, Nagai M, Sugawara Y, Nitta A, Tomata Y, Niu K, Tsuji I. Green tea consumption is associated with lower psychological distress in a general population: the Ohsaki Cohort 2006 Study. Am J Clin Nutr. 2009 Nov;90(5):1390-6. doi: 10.3945/ajcn.2009.28214. Epub 2009 Sep 30. PMID 19793850
- [Background] Wakabayashi C, Numakawa T, Ninomiya M, Chiba S, Kunugi H. Behavioral and molecular evidence for psychotropic effects in L-theanine. Psychopharmacology (Berl). 2012 Feb;219(4):1099-109. doi: 10.1007/s00213-011-2440-z. Epub 2011 Aug 23. PMID 21861094
- [Background] Egashira N, Ishigami N, Pu F, Mishima K, Iwasaki K, Orito K, Oishi R, Fujiwara M. Theanine prevents memory impairment induced by repeated cerebral ischemia in rats. Phytother Res. 2008 Jan;22(1):65-8. doi: 10.1002/ptr.2261. PMID 17705146
- [Background] Lardner AL. Neurobiological effects of the green tea constituent theanine and its potential role in the treatment of psychiatric and neurodegenerative disorders. Nutr Neurosci. 2014 Jul;17(4):145-55. doi: 10.1179/1476830513Y.0000000079. Epub 2013 Nov 26. PMID 23883567
- [Background] Hidese S, Ota M, Wakabayashi C, Noda T, Ozawa H, Okubo T, Kunugi H. Effects of chronic l-theanine administration in patients with major depressive disorder: an open-label study. Acta Neuropsychiatr. 2017 Apr;29(2):72-79. doi: 10.1017/neu.2016.33. Epub 2016 Jul 11. PMID 27396868
- [Background] Paulus W, Classen J, Cohen LG, Large CH, Di Lazzaro V, Nitsche M, Pascual-Leone A, Rosenow F, Rothwell JC, Ziemann U. State of the art: Pharmacologic effects on cortical excitability measures tested by transcranial magnetic stimulation. Brain Stimul. 2008 Jul;1(3):151-63. doi: 10.1016/j.brs.2008.06.002. Epub 2008 Jun 30. PMID 20633382
- [Background] Radhu N, de Jesus DR, Ravindran LN, Zanjani A, Fitzgerald PB, Daskalakis ZJ. A meta-analysis of cortical inhibition and excitability using transcranial magnetic stimulation in psychiatric disorders. Clin Neurophysiol. 2013 Jul;124(7):1309-20. doi: 10.1016/j.clinph.2013.01.014. Epub 2013 Feb 26. PMID 23485366
- [Background] Bajbouj M, Lisanby SH, Lang UE, Danker-Hopfe H, Heuser I, Neu P. Evidence for impaired cortical inhibition in patients with unipolar major depression. Biol Psychiatry. 2006 Mar 1;59(5):395-400. doi: 10.1016/j.biopsych.2005.07.036. Epub 2005 Sep 28. PMID 16197927
- [Background] Lefaucheur JP, Lucas B, Andraud F, Hogrel JY, Bellivier F, Del Cul A, Rousseva A, Leboyer M, Paillere-Martinot ML. Inter-hemispheric asymmetry of motor corticospinal excitability in major depression studied by transcranial magnetic stimulation. J Psychiatr Res. 2008 Apr;42(5):389-98. doi: 10.1016/j.jpsychires.2007.03.001. Epub 2007 Apr 20. PMID 17449060
- [Background] Levinson AJ, Fitzgerald PB, Favalli G, Blumberger DM, Daigle M, Daskalakis ZJ. Evidence of cortical inhibitory deficits in major depressive disorder. Biol Psychiatry. 2010 Mar 1;67(5):458-64. doi: 10.1016/j.biopsych.2009.09.025. Epub 2009 Nov 17. PMID 19922906
- [Background] Jeng JS, Li CT, Lin HC, Tsai SJ, Bai YM, Su TP, Chang YW, Cheng CM. Antidepressant-resistant depression is characterized by reduced short- and long-interval cortical inhibition. Psychol Med. 2020 Jun;50(8):1285-1291. doi: 10.1017/S0033291719001223. Epub 2019 Jun 3. PMID 31155020
- [Background] Ziemann U, Chen R, Cohen LG, Hallett M. Dextromethorphan decreases the excitability of the human motor cortex. Neurology. 1998 Nov;51(5):1320-4. doi: 10.1212/wnl.51.5.1320. PMID 9818853
- [Background] Schwenkreis P, Witscher K, Janssen F, Addo A, Dertwinkel R, Zenz M, Malin JP, Tegenthoff M. Influence of the N-methyl-D-aspartate antagonist memantine on human motor cortex excitability. Neurosci Lett. 1999 Aug 6;270(3):137-40. doi: 10.1016/s0304-3940(99)00492-9. PMID 10462113
- [Background] Di Lazzaro V, Oliviero A, Saturno E, Dileone M, Pilato F, Nardone R, Ranieri F, Musumeci G, Fiorilla T, Tonali P. Effects of lorazepam on short latency afferent inhibition and short latency intracortical inhibition in humans. J Physiol. 2005 Apr 15;564(Pt 2):661-8. doi: 10.1113/jphysiol.2004.061747. Epub 2005 Feb 17. PMID 15718269
- [Background] Ritsner MS, Miodownik C, Ratner Y, Shleifer T, Mar M, Pintov L, Lerner V. L-theanine relieves positive, activation, and anxiety symptoms in patients with schizophrenia and schizoaffective disorder: an 8-week, randomized, double-blind, placebo-controlled, 2-center study. J Clin Psychiatry. 2011 Jan;72(1):34-42. doi: 10.4088/JCP.09m05324gre. Epub 2010 Nov 30. PMID 21208586
- [Background] Borzelleca JF, Peters D, Hall W. A 13-week dietary toxicity and toxicokinetic study with l-theanine in rats. Food Chem Toxicol. 2006 Jul;44(7):1158-66. doi: 10.1016/j.fct.2006.03.014. Epub 2006 Apr 26. PMID 16759779
- [Background] Taylor JJ, Borckardt JJ, George MS. Endogenous opioids mediate left dorsolateral prefrontal cortex rTMS-induced analgesia. Pain. 2012 Jun;153(6):1219-1225. doi: 10.1016/j.pain.2012.02.030. Epub 2012 Mar 22. PMID 22444187
- [Background] Health Quality Ontario. Repetitive Transcranial Magnetic Stimulation for Treatment-Resistant Depression: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Ont Health Technol Assess Ser. 2016 Mar 1;16(5):1-66. eCollection 2016. PMID 27099642
- [Background] Carpenter LL, Janicak PG, Aaronson ST, Boyadjis T, Brock DG, Cook IA, Dunner DL, Lanocha K, Solvason HB, Demitrack MA. Transcranial magnetic stimulation (TMS) for major depression: a multisite, naturalistic, observational study of acute treatment outcomes in clinical practice. Depress Anxiety. 2012 Jul;29(7):587-96. doi: 10.1002/da.21969. Epub 2012 Jun 11. PMID 22689344
- [Background] Levkovitz Y, Isserles M, Padberg F, Lisanby SH, Bystritsky A, Xia G, Tendler A, Daskalakis ZJ, Winston JL, Dannon P, Hafez HM, Reti IM, Morales OG, Schlaepfer TE, Hollander E, Berman JA, Husain MM, Sofer U, Stein A, Adler S, Deutsch L, Deutsch F, Roth Y, George MS, Zangen A. Efficacy and safety of deep transcranial magnetic stimulation for major depression: a prospective multicenter randomized controlled trial. World Psychiatry. 2015 Feb;14(1):64-73. doi: 10.1002/wps.20199. PMID 25655160
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] McClintock SM, Reti IM, Carpenter LL, McDonald WM, Dubin M, Taylor SF, Cook IA, O'Reardon J, Husain MM, Wall C, Krystal AD, Sampson SM, Morales O, Nelson BG, Latoussakis V, George MS, Lisanby SH; National Network of Depression Centers rTMS Task Group; American Psychiatric Association Council on Research Task Force on Novel Biomarkers and Treatments. Consensus Recommendations for the Clinical Application of Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Depression. J Clin Psychiatry. 2018 Jan/Feb;79(1):16cs10905. doi: 10.4088/JCP.16cs10905. PMID 28541649
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Background] Gomez-Ramirez M, Kelly SP, Montesi JL, Foxe JJ. The effects of L-theanine on alpha-band oscillatory brain activity during a visuo-spatial attention task. Brain Topogr. 2009 Jun;22(1):44-51. doi: 10.1007/s10548-008-0068-z. Epub 2008 Oct 9. PMID 18841456
- [Background] Gomez-Ramirez M, Higgins BA, Rycroft JA, Owen GN, Mahoney J, Shpaner M, Foxe JJ. The deployment of intersensory selective attention: a high-density electrical mapping study of the effects of theanine. Clin Neuropharmacol. 2007 Jan-Feb;30(1):25-38. doi: 10.1097/01.WNF.0000240940.13876.17. PMID 17272967
- [Derived] Yuan S, Brown JC, Gold M, Tirrell E, Jones RN, Carpenter LL. Effects of single-dose L-theanine on motor cortex excitability. Clin Neurophysiol. 2021 Sep;132(9):2062-2064. doi: 10.1016/j.clinph.2021.07.003. Epub 2021 Jul 10. No abstract available. PMID 34293527

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We screened and enrolled 11 subjects altogether. 10 subjects in total completed the study. As this is a cross-over study, so each arm has 10 subjects.
Groups:
- L-Theanine First, Then Placebo: Subject will receive 400mg single dose of L-theanine, by oral ingestion with water. The capsules are prepared and dispensed by hospital pharmacy, with the investigator and participant both blinded.
  L-theanine: The subject will receive paired-pulse TMS (ppTMS) procedure before and 30min after taking the drug orally, to assess motor cortex excitability, measured by surface electromyogram (EMG). The ppTMS procedure is administered by a TMS stimulator controlled a software named Signal. The coil of the stimulator is placed above the scalp where the stimulation would activate the left primary motor cortex region that controls the right thumb. When a pulse is delivered by the coil, the EMG over a thumb muscle (abductor pollicis brevis) will record a motor-evoked potential on the tracing. Cross-over with placebo in two separate sessions at least 72 hours apart.
  Placebo: The subject will receive ppTMS procedure before and 30min after taking the drug orally, to assess motor cortex excitability, measured by surface electromyogram (EMG). The ppTMS procedure is administered by a TMS stimulator controlled a software named Signal. The coil of the stimulator is placed above the scalp where the stimulation would activate the left primary motor cortex region that controls the right thumb. When a pulse is delivered, the EMG over the abductor pollicis brevis will record a motor-evoked potential on the tracing. Cross-over with L-theanine in two separate sessions at least 72 hours apart.
- Placebo First, Then L-Theanine: Subject will receive 400mg single dose of matching Placebo, by oral ingestion with water. The capsules are prepared and dispensed by hospital pharmacy, with the investigator and participant both blinded.
  L-theanine: The subject will receive paired-pulse TMS (ppTMS) procedure before and 30min after taking the drug orally, to assess motor cortex excitability, measured by surface electromyogram (EMG). The ppTMS procedure is administered by a TMS stimulator controlled a software named Signal. The coil of the stimulator is placed above the scalp where the stimulation would activate the left primary motor cortex region that controls the right thumb. When a pulse is delivered by the coil, the EMG over a thumb muscle (abductor pollicis brevis) will record a motor-evoked potential on the tracing. Cross-over with placebo in two separate sessions at least 72 hours apart.
  Placebo: The subject will receive ppTMS procedure before and 30min after taking the drug orally, to assess motor cortex excitability, measured by surface EMG. The ppTMS procedure is administered by a TMS stimulator controlled a software named Signal. The coil of the stimulator is placed above the scalp where the stimulation would activate the left primary motor cortex region that controls the right thumb. When a pulse is delivered by the coil, the EMG over the abductor pollicis brevis will record a motor-evoked potential on the tracing. Cross-over with L-theanine in two separate sessions at least 72 hours apart.
Period: Overall Study
Arm/Group | L-Theanine First, Then Placebo | Placebo First, Then L-Theanine
Started | 5 | 6
First Intervention | 4 | 6
Washout (72 hours at least) | 4 | 6
Second Intervention | 4 | 6
Completed | 4 | 6
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: This is a cross-over study, therefore, the total number of subjects is 10.
Groups:
- L-Theanine and Placebo Cross-over in All Subjects: Subject will receive 400mg single dose of L-theanine or Placebo, by oral ingestion with water. After 72 hours washout period, the same subject will then receive 400mg single dose of Placebo or L-theanine (opposite condition from the first dose). The capsules are prepared and dispensed by hospital pharmacy, with the investigator and participant both blinded. All subjects receive both conditions of drugs.
Arm/Group | L-Theanine and Placebo Cross-over in All Subjects
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.7 (3.1)
Handedness (Right) [Count of Participants; unit: Participants] | 10
Multilingual [Count of Participants; unit: Participants] | 3
Years of Education [Mean (Standard Deviation); unit: years] | 20.8 (2.4)
Average Sleep Hours [Mean (Standard Deviation); unit: Hours] | 7.4 (0.6)
Daily Coffee Drinker [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: The Change of Motor Cortex Excitability Measures by ppTMS
Description: The changes of Short-interval Intracortical Inhibition (SICI), Intracortical Facilitation (ICF), and Long-interval Intracortical Inhibition (LICI) before and 30 minutes after each drug administration.
  SICI, ICF and LICI are paired-pulse TMS (ppTMS)-EMG outcome measures that assess the activity of motor cortex GABA-A, NMDA and GABA-B interneurons, respectively. They are measured by the ratio between the peak-to-peak amplitude of motor-evoked potential (MEP) elicited by a testing TMS pulse (120% of the intensity of the resting motor threshold, following a conditioning pulse at different inter-stimuli interval, 2-5 milliseconds for SICI, 10-20 milliseconds for ICF, 100-200 milliseconds for LICI) and the peak-to-peak MEP amplitude elicited by a single pulse (120% of the intensity of the resting motor threshold).
  The baseline-to-post-drug change of SICI, ICF and LICI elicited by L-theanine will be compared to that elicited by placebo within each subject.
Time Frame: Before and 30 minutes after each drug administration (no long-term follow up as this is a study on acute effect of a single-dose agent).
Population: This is a cross-over study, therefore each subject will receive the drug conditions in both arms. The outcomes will be compared using Wilcoxon Signed-rank test to see if L-theanine elicits different changes of SICI, ICF or LICI within each individual than placebo does.
Measure: Mean (Standard Error); unit: Ratio
Groups:
- L-Theanine: Subject will receive 400mg single dose of L-theanine, by oral ingestion with water. The capsules are prepared and dispensed by hospital pharmacy, with the investigator and participant both blinded.
  The baseline-to-post-drug change of SICI, ICF and LICI elicited by L-theanine will be compared to that elicited by placebo within each subject.
- Placebo: Subject will receive 400mg single dose of matching Placebo, by oral ingestion with water. The capsules are prepared and dispensed by hospital pharmacy, with the investigator and participant both blinded.
  The baseline-to-post-drug change of SICI, ICF and LICI elicited by L-theanine will be compared to that elicited by placebo within each subject.
Arm/Group | L-Theanine | Placebo
Number analyzed (Participants) | 10 | 10
Ratio
  SICI | 0.059 (0.028) | 0.005 (0.060)
  ICF | 0.073 (0.073) | -0.341 (0.176)
  LICI | 0.145 (0.100) | -0.068 (0.053)

2. Secondary Outcome: The Change of Visual Analog Scale (VAS)
Description: VAS is a quick scale to assess and track how the participant subjectively feels through out each study session, e.g. anxiety, depression, excitement, etc. The score for each word ranges from "0" being the least in your life and "100" being the most in your life. It takes 3-4 minutes to complete each VAS, and there are 4 takes of VAS during each session. The outcome measure is the change of VAS throughout the 4 time points: 1) before the baseline ppTMS procedure; 2) before drug administration; 3) 30 minutes after drug administration; 4) before discharge from the session, during the session.
Time Frame: Throughout each session; each session lasts up to 3 hours; 2 sessions for each subject. The 2 sessions are 3-7 days apart.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 72 hours after administration of each drug condition (single dose of L-theanine or placebo).
Arm/Group | L-Theanine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/11 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-Theanine (N=11) | Placebo (N=11)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) — This was associated with the testing method (transcranial magnetic stimulation) before data collection. The subject recovered back to baseline mental status quickly from the syncope and did not need emergent medical care or hospitalization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT04749745/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT04749745/ICF_001.pdf